CLINICAL TRIAL: NCT06930053
Title: Effect of Action Observation Training Versus Core Stability Training on Hand Functions in Children With Hemiplegic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ahmed Abdou Ragab Abdou, Demonstrator, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KFSIRB200-325
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Hand Functions on Hemiplegic Cerebral Palsy
Keywords: Action observation training (AOT)

STUDY DESIGN:
Intervention Model Description: Treatment protocol in Group A, Core stability training:
  The study group will receive core stability exercises, which consist of three levels. Each level took 4 weeks. The difficulty of each level varies in proprioception, balance, and stability as it started from exercising on a stable surface "mat" and ended with unstable surface "physioball" .
  Treatment protocol in Group B, Action observation therapy protocol:
  The examined group got 30 minutes of a standard,selected physical therapy program in addition to 30 minutes of AOT on the upper limb (total session time: 1 hour), 3 sessions per week for three consecutive months (total therapy time: 3 hours/week). Action observation was executed with therapist guidance and repeated practice (3 repetitions for each task).
  Treatment protocol in Group c, combination of Action observation therapy and core stability training
Who Masked: Participant
Masking Description: The participants will not know the details of the intervention of the other groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment protocol in Group A, Core stability training (Active Comparator): The study group will receive core stability exercises, which consist of three levels. Each level took 4 weeks. The difficulty of each level varies in proprioception, balance, and stability as it started from exercising on a stable surface "mat" and ended with unstable surface "physioball". The first simple level involves supine abdominal draw (3 sets per 20 repetitions), abdominal draw-in with a double knee to chest (3 sets/20 repetitions), and supine twist (3 sets per 20 repetitions). The second medium level involves pelvic bridging (3 sets per 3-5 repetitions) and twists with a medicine ball (3 sets per 10-20 repetitions). The third difficult level involves bridging with head-on physioball holding this position for 3-5 seconds, then slowly relaxing (3 sets per 10-20 repetitions), and prone bridging (3 sets per 3-repetitions). There was a 30-second rest between sets . The program will be applied 30 minutes a day for 3 days a week for 12 weeks. in addition to 30 minutes of a standar
  Interventions: Other: Core stability training
- Group B, Action observation therapy (Active Comparator): The examined group got 30 minutes of a standard,selected physical therapy program in addition to 30 minutes of AOT on the upper limb (total session time: 1 hour), 3 sessions per week for three consecutive months (total therapy time: 3 hours/week). Action observation was executed with therapist guidance and repeated practice (3 repetitions for each task). The child has been requested to perform the watched task with the same tool after observing a 3-minute video for each task on an adjustable monitor screen positioned one meter infront of him or her from forward, sideways, and backward directions. The therapist sat beside the child to provide verbal comments during the excursion and to guide the child's movement
  Interventions: Other: Action observation therapy
- Group c, combination of Action observation therapy and core stability training . (Active Comparator): Group c, combination of Action observation therapy and core stability training .
  Interventions: Other: combination of Action observation therapy and core stability training .

INTERVENTIONS:
Other: Core stability training — The study group will receive core stability exercises, which consist of three levels. Each level took 4 weeks. The difficulty of each level varies in proprioception, balance, and stability as it started from exercising on a stable surface "mat" and ended with unstable surface "physioball". The first simple level involves supine abdominal draw (3 sets per 20 repetitions), abdominal draw-in with a double knee to chest (3 sets/20 repetitions), and supine twist (3 sets per 20 repetitions). The second medium level involves pelvic bridging (3 sets per 3-5 repetitions) and twists with a medicine ball (3 sets per 10-20 repetitions). The third difficult level involves bridging with head-on physioball holding this position for 3-5 seconds, then slowly relaxing (3 sets per 10-20 repetitions), and prone bridging (3 sets per 3-repetitions). There was a 30-second rest between sets . The program will be applied 30 minutes a day for 3 days a week for 12 weeks. in addition to 30 minutes of a standard
  Arms: Treatment protocol in Group A, Core stability training
Other: Action observation therapy — The examined group got 30 minutes of a standard,selected physical therapy program in addition to 30 minutes of AOT on the upper limb (total session time: 1 hour), 3 sessions per week for three consecutive months (total therapy time: 3 hours/week). Action observation was executed with therapist guidance and repeated practice (3 repetitions for each task). The child has been requested to perform the watched task with the same tool after observing a 3-minute video for each task on an adjustable monitor screen positioned one meter infront of him or her from forward, sideways, and backward directions. The therapist sat beside the child to provide verbal comments during the excursion and to guide the child's movement.The AOT for the examined group included six unimanual tasks and six bimanual tasks. The unimanual tasks included pressing a rubber stamp, stacking cups, drinking water from a cup, grabbing a pen, flipping cards, and putting things on a stick. The bimanual tasks were opening a bo
  Arms: Group B, Action observation therapy
Other: combination of Action observation therapy and core stability training . — combination of Action observation therapy and core stability training .
  Arms: Group c, combination of Action observation therapy and core stability training .

SUMMARY:
This study will be conducted to compare between the effectiveness of Action observation therapy (AOT) and core stability training and the combination of Action observation therapy (AOT) and core stability training on hand function in hemiplegic CP

DETAILED DESCRIPTION:
Cerebral palsy (CP) refers to a collection of permanent mobility and postural impairments that are caused by non-progressive disruptions in the fetal or infant brain throughout development. Children with CP have motor abnormalities that are commonly accompanied by sensory and cognition disorders as well as seizures and secondary musculoskeletal difficulties. Cerebral palsy can be broken down into four basic categories based on the degree of activity restriction: motor abnormalities, accompanying impairments, anatomical and neuroimaging results, and etiology and timing of motor problems . It is a chronic and disabling childhood condition that occurs in 1.5/1,000 to 3/1,000 live births .Pregnancy age under 20 years, birth weight under 2500 gramme , risk factors related to the mother, pregnancy variables (placental dislodgement ,twining), and fetal factors are all examples of CP causes or risk factors(bradycardia, fetal malformation, poor fetal growth) As a well-known neurodevelopmental disorder, CP can begin in early childhood and last throughout life. For example, non-progressive abnormalities in the growing fetus or infant brain might cause activity limitations, poor sensation and cognition as well as mobility and posture issues .

Three out of every 1000 children with CP have a movement and coordination disorders which are compromised in people with CP due to both decreased brain control and secondary alterations in muscle characteristics. It is difficult to quantify the degree and functional significance of changes in muscle characteristics for individual patients with CP, which makes therapy planning difficult .

Early intervention for the upper limb in hemiplegia remains challenging, though progress is being made. It was concluded that the difficulties of outcome assessment in the youngest infants and children, which make evaluation of interventions very difficult. The diversity of the population under study, in terms of lesion type, differences in post-lesional reorganization, and the degree to which other factors such as vision, sensation, and cognitive ability impact on hand function, must also be considered .

ELIGIBILITY:
Inclusion Criteria:

1. Their age will be ranged from four to eight years.
2. Their grade of spasticity will be from 1 to 1+ according to Modified Ashworth scale .
3. They will be on Level I and II according to Gross Motor Functional Classification System (GMFCS) .
4. The child will be able to follow verbal commands and instructions.

Exclusion Criteria:

- The children will be excluded if they have one of the following:

1. history of orthopedic surgery in the affected upper limb
2. Botox injection in the upper limb in the past 6 months or planned to have one during study time

4-Fixed deformities or contructures in spine. 5- A history of epileptic seizure and cardiac or respiratory problems. 6- Severe hearing and visual defect.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2025-05-09 (Actual); Primary Completion 2025-08-09 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
evaluates the quality of upper extremity skill function through 33 activity items of 4 domains: dissociated movement consists of 19 items, grasp consists of 6 items, weight-bearing consists of 5 items, and protective extension consists of 3 items | After 12 week
  The Quality Upper Extremity Skill Test (QUEST)
Assessment of the grip strength | After 12 week
  Assessment of the grip strength by using Hand and Held Dynamometer:
Measure hand function for activities of daily living. It has 7 items include: writing, turning over 3-by-5 inch cards, picking up small common objects, simulated feeding, stacking checkers, picking up large light objects and picking up large heavy object | After 12 week
  Jebsen Hand Function Test

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Bedair Ibrahim, Professor of Physical Therapy, Principal Investigator — kafr-elsheikh university
Locations (1):
- Ahmed Abdou Ragab Abdou, Beheira, Egypt

IPD SHARING:
Plan to Share IPD: No